CLINICAL TRIAL: NCT01685970
Title: Comparison of Using the Same-day 2 Sachets Picosulfate Versus High Volume PEG Bowel Preparation for Afternoon Colonoscopy
Brief Title: Comparison of Same-day 2 Sachets Picosulfate Versus High Volume PEG for Afternoon Colonoscopy
Acronym: SP2HP
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Inje University (Other)
Responsible Party: Principal Investigator, Eun Hee Seo, MD, Comparison of using the same-day 2 sachets picosulfate versus high volume PEG bowel preparation for aternoon colonoscopy, Inje University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: HGI-2012-09
Record Dates: First submitted 2012-09-12; First posted 2012-09-17 (Estimated); Last update posted 2012-09-17 (Estimated); Status verified 2012-09

CONDITIONS: Colonoscopy
Keywords: Bowel preparation; colonoscopy; polyethylene glycol; picosulfate
MeSH Terms: interventions — picosulfate sodium

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High volume Split-dose PEG (Placebo Comparator): Patients who are scheduled afternoon colonoscopy ingest high volume split-dose PEG for bowel preparation
  Interventions: Drug: High volume split-dose PEG
- 2 sachets of picosulfate (Active Comparator): Patients who are scheduled afternoon colonoscopy ingest 2 sachets of picosulfate at the day of colonoscopy.
  Interventions: Drug: 2 sachets of picosulfate

INTERVENTIONS:
Drug: High volume split-dose PEG — High volume split-dose PEG 2L/2L 2 times before the day and at the day of colonoscopy
  Other Names: Polyethylene glycol(Colyte)
  Arms: High volume Split-dose PEG
Drug: 2 sachets of picosulfate — 2 sachets of picosulfate 2 times for bowel preparation at the day of colonoscopy
  Other Names: sodium picosulfate
  Arms: 2 sachets of picosulfate

SUMMARY:
Comparison of using the same-day 2 sachets picosulfate versus high volume PEG bowel preparation for afternoon colonoscopy Morning only same-day 2 sachets picosulfate may enhance patient tolerability and have similar bowel cleansing efficacy compared to standard method using high volume split-dose PEG.

The investigators aimed to evaluate the efficacy and tolerability of bowel preparation protocols with same-day 2 sachets picosulfate compared to conventional high volume (4L) split-dose for afternoon colonoscopy.

DETAILED DESCRIPTION:
Split-dose PEG (4L) regimens is a standard regimen for bowel preparation because it has better preparation quality and tolerability than single dose 4L PEG regimens. However, although patients drink each 2L separately, the total volume of 4 L PEG is still quite burdensome volume to ingest. In addition, in split dose method, night dose of day before the procedure make patient to suffer from sleep disturbance because of frequent diarrhea and abdominal discomfort.

The investigators aimed to evaluate the efficacy and tolerability of bowel preparation protocols with same-day 2 sachets picosulfate compared to conventional high volume (4L) split-dose for afternoon colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Adult outpatients who undergo afternoon colonoscopy for screening, surveillance or with symptoms

Exclusion Criteria:

* pregnancy,
* breast feeding,
* prior history of surgical large bowel resection,
* severe medical condition such as severe cardiac,
* hepatic, or
* renal failure (creatinine ≥ 3.0 mg/dL (normal 0.8-1.4 mg/dL)),
* significant gastric paresis or gastric outlet obstruction or ileus,
* known or suspected bowel obstruction or perforation,
* drug addiction or major psychiatric illness,
* allergy to PEG and refusal to participate in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-09; Primary Completion 2012-11 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Quality of bowel preparation | 3 months
  Quality of bowel preparation using Ottawa bowel preparation scale

SECONDARY OUTCOMES:
Tolerability | 3 months
  Tolerability of bowel preparation regimen is assessed by patient questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Tae Oh Kim, Ph D, Study Director — Haeundae Paik Hospital, Inje University College of Medicine
Locations (1):
- Haeundae Paik Hospital, Inje University College of Medicine, Busan, South Korea